CLINICAL TRIAL: NCT03382288
Title: Clinical Trial ES 900 - 2016
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haag-Streit AG (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1023191
Record Dates: First submitted 2017-11-10; First posted 2017-12-22 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Optical Biometry of the Human Eye; General Analysis of the Anterior Chamber of the Human Eye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Examination of participants (Experimental): Examination of participants by means of the investigational device, Eyestar 900 as well as the comparative devices.
  Interventions: Device: EYESTAR 900

INTERVENTIONS:
Device: EYESTAR 900 — EYESTAR 900 is an optical biometry device used to create a geometrical representation of the eye by means of optical interferometry. The experimental intervention is an optical, non-contact examination with the investigational device EYESTAR 900.

SUMMARY:
The primary objective of this clinical trial is to assess the clinical performance of the investigational device. To that end, for each measure and the in-vivo repeatability will be quantified, as well as the mean measurement deviation with respect to the current gold standard device. As a secondary objective of the study, raw measurement data will be collected, to allow for improvements of existing algorithms, development of additional measure and and for retrospective analysis.

DETAILED DESCRIPTION:
EYESTAR 900 (the investigational device) is a new device by HAAG-STREIT AG, for measurement of optical biometry and advanced corneal topography by swept-source optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* volunteers with phakic eyes, no cataract surgery indicated and with existing vitreous;
* patients seeking cataract surgery;
* patients with pseudophakic eye;
* patients with oil-filled eye;
* patients with aphakic eye.

Exclusion Criteria:

* underage patients (younger than 18 years);
* vulnerable patients;
* inability to give informed consent;
* inability to maintain stable fixation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Keratometry-Measurands | Through study completion, approximately 9 months.
  In-vivo repeatability and confidence interval of mean deviation with respect to comparator device, for K1, K2 (R1, R2, AST) in [dpt]; Axis in [°].
Axial measurands | Through study completion, approximately 9 months
  In-vivo repeatability and confidence interval of mean deviation with respect to comparator device, for CCT in [µm]; AD in [mm]; ACD in [mm]; LT in [mm]; AL in [mm].
Imaging | Through study completion, approximately 9 months
  In-vivo repeatability and confidence interval of mean deviation with respect to comparator device, for WTW in [mm]; ICX, ICY in [mm]; PD in [mm]; PCX, PCY in [mm].
Anterior corneal topography | Through study completion, approximately 9 months
  In-vivo repeatability and confidence interval of mean deviation with respect to comparator device, for elevation in [µm ]; axial curvature in [dpt].
Posterior corneal topography | Through study completion, approximately 9 months
  In-vivo repeatability and confidence interval of mean deviation with respect to comparator device, for elevation in [µm]; axial curvature in [dpt].
Corneal pachymetry | Through study completion, approximately 9 months
  In-vivo repeatability and confidence interval of mean deviation with respect to comparator device, for CT in [µm ].
Posterior corneal keratometry | Through study completion, approximately 9 months
  In-vivo repeatability and confidence interval of mean deviation with respect to comparator device, for PK1, PK2 (PR1, PR2, PAST) in [dpt]; PAxis in [°].

SECONDARY OUTCOMES:
Aquisition of volumetric OCT Data of the eye. | Through study completion, approximately 9 months
  Data is collected, but not processed within the scope of this clinical trial.
Aquisition of photographic images of the eye. | Through study completion, approximately 9 months
  Data is collected, but not processed within the scope of this clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: David Goldblum, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland